CLINICAL TRIAL: NCT06989840
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of TVB-3567 in Healthy Participants With or Without Acne and to Assess the Effect of Food in Healthy Participants
Brief Title: Phase 1 Study to Evaluate the Safety, Tolerability, PK, and PD of TVB-3567 in Healthy Participants With or Without Acne
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sagimet Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SB3567-CLIN-001
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A (SAD in Healthy Participants) (Experimental)
  Interventions: Drug: TVB-3567; Drug: Placebo
- Part B (Food Effect) (Experimental)
  Interventions: Drug: TVB-3567
- Part C (MAD in Healthy Participants) (Experimental)
  Interventions: Drug: TVB-3567; Drug: Placebo
- Part D (MAD in Acne Participants) (Experimental)
  Interventions: Drug: TVB-3567; Drug: Placebo

INTERVENTIONS:
Drug: TVB-3567 — Orally administered capsule
Drug: Placebo — Orally administered capsule
  Arms: Part A (SAD in Healthy Participants); Part C (MAD in Healthy Participants); Part D (MAD in Acne Participants)

SUMMARY:
This is a 4-part study. Part A will be a randomized, double-blind, placebo-controlled investigation of single ascending doses (SAD) to assess the safety, tolerability, pharmacokinetics (PK), and pharmacodynamic (PD) biomarkers of TVB-3567 administered orally in healthy participants. Part B will be a randomized, open-label, 2-way crossover investigation to assess the effect of food on a single dose TVB-3567 administered orally in healthy participants. Parts C and D will be randomized, double-blind, placebo-controlled investigations of multiple ascending doses (MAD) to assess the safety, tolerability, PK, and PD/biomarkers of TVB-3567 administered orally in healthy participants without and with moderate to severe acne, respectively.

ELIGIBILITY:
Inclusion Criteria:

Healthy Participants (Parts A, B and C)

1. Healthy, adult, male or female 18-55 years of age
2. Body mass index (BMI) ≥18.0 and ≤32.0 kg/m2
3. Medically healthy with no clinically significant medical history
4. Understands the study procedures in the informed consent form (ICF) and willing and able to comply with the protocol

Healthy Participants with Acne (Part D only)

Participants must meet all of the above criteria, as well as the following inclusion criteria to be eligible for participation in the study:

1. BMI ≥18.0 and ≤37.0 kg/m2.
2. Must be diagnosed with moderate to severe acne vulgaris

Exclusion Criteria:

Healthy Participants (Parts A, B and C)

1. History or presence of clinically significant medical or psychiatric condition or disease
2. History or presence of hypersensitivity or idiosyncratic reaction to the study drug or related compounds including over the counter acne products.
3. Has a clinically significant ophthalmic examination finding
4. Female participant of childbearing potential
5. Unable to refrain from or anticipates the use of:

   * Any drugs, including prescription and non-prescription medications, herbal remedies, or vitamin supplements
   * Any topical anti-acne treatment on the face
   * Any drugs known to be moderate or strong inducers of CYP3A4 enzymes, BCRP, and/or P gp, including St. John's Wort, beginning 28 days prior to the first dosing.
   * Part C only: Any previous tretinoin treatments, including tazarotene, adapalene, isotretinoin, and all-trans retinoic acid.

Healthy Participants with Acne (Part D only)

Participants must not be enrolled if they do not meet any of the above criteria, as well as the following exclusion criteria:

1. Unable to refrain from or anticipates the use of:

   * Any previous tretinoin treatments, including tazarotene, adapalene, isotretinoin, and all trans retinoic acid.
   * Photoelectric therapy, dermabrasion, or chemical peeling
   * Intra-articular and systemic corticosteroid therapy
2. Significant skin diseases

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Part A - Incidence of adverse events (AEs) and serious adverse events (SAEs) | Baseline to 7 to 8 days after dosing
Part B - Plasma AUC0-t in fasted and fed conditions | Baseline to Day 4
  Area under the concentration-time curve from time zero until the last observed concentration
Part B - Plasma AUC0-inf in fasted and fed conditions | Baseline to Day 4
  Area under the concentration-time curve from time zero to infinity
Part B - Plasma Cmax in fasted and fed conditions | Baseline to Day 4
  Maximum concentration measurement in plasma
Part B - Incidence of adverse events (AEs) and serious adverse events (SAEs) under fasted and fed conditions | Baseline to 7 to 8 days after dosing
Part C - Incidence of adverse events (AEs) and serious adverse events (SAEs) | Baseline to 13 to 15 days after the last dose
Part D - Incidence of adverse events (AEs) and serious adverse events (SAEs) | Baseline to 13 to 15 days after the last dose

CONTACTS AND LOCATIONS:
Locations (2):
- Celerion, Inc., Tempe, Arizona, United States
- Nucleus Network, Melbourne, Victoria, Australia